CLINICAL TRIAL: NCT00416962
Title: An Open-Label, Multiple Dose, Randomized, Three-Period Crossover Study in Healthy Volunteers to Evaluate the Effect of co-Administration of Amantadine 100 mg BID and Oseltamivir 75 mg BID on the Pharmacokinetic Properties of Amantadine and Oseltamivir.
Brief Title: Safety and Pharmacokinetic Effects of Oseltamivir Alone or in Combination With Amantadine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CSYO380A2101
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2007-11-30 (Estimated); Status verified 2007-11

CONDITIONS: Healthy
Keywords: Oseltamivir, amantidine, Symmetrel, Tamiflu
MeSH Terms: interventions — Amantadine; Oseltamivir

INTERVENTIONS:
Drug: amantadine hydrochloride
Drug: oseltamivir phosphate

SUMMARY:
This study is designed to assess the safety and pharmacokinetic effects of oseltamivir administration alone or in combination with amantadine in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects aged 18 to 45 years, and in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests
* Vital signs within the following ranges:

  * oral body temperature 35.0 - 37.5°C
  * systolic blood pressure 90 - 140 mm Hg
  * diastolic blood pressure 50 - 90 mm Hg
  * pulse rate 40 - 90 bpm
* Female subjects of child bearing potential must be using double-barrier local contraception (for example, intra-uterine device plus condom, or spermicidal gel plus condom) or have been surgically sterilized at least 6 months prior before study start, with supportive clinical documentation OR Postmenopausal women must have no regular menstrual bleeding for at least 1 year prior to inclusion.
* Body mass index must be within 18 - 30 kg/m2. Subjects must weigh at least 50 kg.

Exclusion Criteria:

* Smokers (use of tobacco products in the previous 3 months). Smokers will be defined as those who report tobacco use or have a urine cotinine greater than 500 ng/mL
* Female subjects who are pregnant or lactating
* Participation in any clinical investigation involving medical intervention within 4 week prior to study start.
* Donation or loss of ≥ 400 mL of blood within 8 weeks prior to study start, or longer if required by local regulation.
* Significant illness within 2 weeks before study start.
* A past personal or close family medical history of clinically significant ECG abnormalities or of a prolonged QT-interval syndrome.
* History of autonomic dysfunction (for example, history of fainting).
* History of acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease, treated or untreated),
* History of clinically significant drug allergy or history of atopic allergy (asthma, urticaria, eczematous dermatitis). A known hypersensitivity to the study drug or to similar drugs.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs, or which may jeopardize the subject in case of participation in the study, including bowel, gastrointestinal, renal, pancreatic, hepatic, hematological, immunological, or neurological disorders.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18
Dates: Start 2006-08; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To characterize the pharmacokinetics of amantadine following twice daily administration alone or in combination with twice daily oseltamivir in healthy volunteers.
To characterize the pharmacokinetics of oseltamivir following twice daily administration alone or in combination with twice daily amantadine in healthy volunteers.

SECONDARY OUTCOMES:
To assess the safety and tolerability of twice daily oseltamivir and twice daily amantadine when given alone and when given in combination.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigator site
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Morrison D, Roy S, Rayner C, Amer A, Howard D, Smith JR, Evans TG. A randomized, crossover study to evaluate the pharmacokinetics of amantadine and oseltamivir administered alone and in combination. PLoS One. 2007 Dec 12;2(12):e1305. doi: 10.1371/journal.pone.0001305. PMID 18074029